CLINICAL TRIAL: NCT06783595
Title: Peri-implant Mucosal Changes Over Time Following Implant Provisional Removal in the Esthetic Zone
Status: Recruiting | Type: Observational
Sponsor: Loma Linda University (Other)
Responsible Party: Sponsor
Other Study IDs: 5230566
Record Dates: First submitted 2025-01-14; First posted 2025-01-20 (Actual); Last update posted 2025-11-19 (Actual); Status verified 2025-11

CONDITIONS: Tooth Loss; Implant Site Reaction
Keywords: immediate implant placement; provisional; impression
MeSH Terms: conditions — Tooth Loss

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Other: intraoral scan — Device that scans the mouth with by taking numerous pictures of the mouth and stitches them together to form a three-dimensional copy of the patient teeth.

SUMMARY:
The study will examine the temporary volumetric change that happens in the gums around an implant crown when the crown is removed. The main question of the study is "how much time has to pass to see a significant change, especially when there could be a need to make a mold of the surrounding gum to make a new crown?"

The area of the implant crown will be scanned with an intra-oral scanner over a period of 15 minutes.

DETAILED DESCRIPTION:
When an implant crown is removed, the gum in the area, usually supported by the crown, might go through temporary changes once that support is gone. While the change itself may be temporary, some ways to make a final crown that would be esthetically pleasing might require making a copy of the temporary crown or a mold of the gum around the crown.

This study will involve the removal of an implant crown at a site where a failing tooth was removed, and a dental implant and a crown was placed into the extraction socket. Once the subject enrolls in the study, the area of the implant crown will be scanned right after the removal of the implant crown, and 1, 2, 3, 5, 7, 10, and 15 minutes after the removal of the crown. In order to record the exact location of the implant, a tag will be placed onto the implant and the tag will be scanned as well. The subject's crown will be also scanned so that all the data can be overlaid on top of each other to assess the actual change that occurs. After, the crown will be re-inserted in the patient's mouth so that the gum can rebound back to its original shape.

If the patient is able to return in the near future for a new crown, the patient will be asked to make one final scan of the mouth to see if there is any changes in the gums between that of the old and the new crown. This will show if the shape of the crown under the gums might have an effect on how the gums might look.

The study will look into whether an immediate change might happen, and how much change actually takes place over the 15 minutes, in whichever direction it might happen.

ELIGIBILITY:
Inclusion Criteria:

* Patient must have a maxillary anterior immediate implant and provisionalization treatment completed.
* The adjacent tooth next to the implant should be a natural tooth
* The temporary crown must have been in place for a minimum of 4 months
* The patient needs to be of general good health, with no significant medical history or social habits that might directly affect the hard and soft tissue
* Patient must have generally good oral hygiene without any history of gum disease or gum recession of other teeth around the region of interest

Exclusion Criteria:

* Patient with an implant crown that has no teeth next to the implant crown
* Patients who have an active gum disease

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients selected for the participation in the study will be solely from the Center of Implant Dentistry at Loma Linda University School of Dentistry.
Sampling Method: Probability Sample
Enrollment: 34 (Estimated)
Dates: Start 2024-04-24 (Actual); Primary Completion 2026-01 (Estimated); Study Completion 2026-02 (Estimated)

PRIMARY OUTCOMES:
Peri-implant mucosal volumetric change | Change between baseline and 15 minutes post initial crown removal
  The mucosal volumetric change will be a composite measurement of the outside and inside portion of the peri-implant gum area by a 3D analyzing software. The 3D image that has been captured from an intra-oral scan will be analyzed during the time interval mentioned in the study description. This measurement is representing the horizontal change, and will be recorded in millimeters (mm). The critical analysis will be placed as changes from 0.5mm. Any change more than 0.5mm will be considered a large amount of change.

SECONDARY OUTCOMES:
Vertical gingival margin discrepancy | Change between baseline and 15 minutes post initial crown removal
  This is the composite measure of the coronal-apical shift of the crown margin once the crown is removed. This would be the vertical change happening when you are looking straight at the subject. The vertical height will be measured from the actual crown margin to the resulting crown margin following crown removal, and the measurement will be recorded as millimeters (mm.) Any change more than 0.5mm will be considered a significant change.

CONTACTS AND LOCATIONS:
Overall Officials: Joseph Kan, DDS, MS, Principal Investigator — Loma Linda University
Locations (1):
- Loma Linda University - Center of Implant Dentistry, Loma Linda, California, United States

IPD SHARING:
Plan to Share IPD: No